CLINICAL TRIAL: NCT00951730
Title: Evaluation of a Simplified Method for Diagnosis of Sleep Apnea in Children and Adults With Down Syndrome
Acronym: SAOS/T21
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0808017; 2008-A01273-52 (Other: AFSSAPS)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Adult; Children; Sleep apnea; Sleep hypopnea; Polysomnography
MeSH Terms: conditions — Down Syndrome; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Down syndrome: Adult and children with Down syndrome.
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — Polysomnography is the method of choice for the diagnosis of sleep apnea. This test lasts for one night in hospital.

SUMMARY:
People with Down syndrome are at increased risk of sleep apnea, not only from obstruction of the upper airway, but also of central origin. According to published data, sleep apnea may occur in at least 40% of children and adults with Down syndrome. Consequences of these sleep apnea are numerous : failure to thrive, cognitive decline, high blood pressure, heart disease, accident due to day sleepiness, fatigue. This condition is treatable in people with Down syndrome, as it is in ordinary people.

Diagnosis of sleep apnea in people with Down syndrome is therefore a major concern. In addition, data regarding age of apparition of this complication are missing, making repeated screening necessary.

Polysomnography is the method of choice for the diagnosis of sleep apnea. Unfortunately, it is time consuming and sleep departments are heavily busy.

DETAILED DESCRIPTION:
The main objective of our study is to evaluate an easier screening strategy combining questionnaire and overnight recording of few data, compared to polysomnography.

We hope our strategy will permit regular screening for people with Down syndrome, helping us to draw guidelines for the survey of sleep apnea in this population.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome
* Patient (or parents of children) affiliated in a Social Regimen
* Written consent signed (by parents for the children)

Exclusion Criteria:

* Severe heart failure
* Insufficient autonomy
* Diagnosis of insanity, or behavioural problems

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Down syndrome
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Apnea / hypopnea events index determined by reading the complete polysomnography (review reference) and apnea / hypopnoea events index determined by the simplified five parameters of the polysomnography | At 15 days after enroling

SECONDARY OUTCOMES:
Questionnaire on sleep | At inclusion and at the end (18 months)
Psychometric tests | At inclusion and at the end (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte De Freminville, MD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - CHU de Grenoble, Grenoble
  - Hospices Civiles de lyon, Lyon
  - CHU de Saint-Etienne, Saint-Etienne